CLINICAL TRIAL: NCT06462677
Title: Surveillance of Emerging Pathogens to Ensure Blood Supply Safety
Status: Withdrawn | Type: Observational
Why Stopped: The kits were FDA and Health Canada approved and therefore the clinical trial is no longer needed.
Sponsor: Canadian Blood Services (Other)
Responsible Party: Principal Investigator, Mindy Goldman, Medical Director - Donation Policy and Studies, Canadian Blood Services
Other Study IDs: Version 02
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Babesioses, Human
MeSH Terms: conditions — Babesiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be collected from the diversion pouch during blood donation and added to a lysis tube which will be used to test for the present of Babesia nucleic acid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Manitoba whole blood donors: All whole blood donors giving blood in Manitoba will be collected for Babesia NAT testing to understand the prevalence of babesiosis in the Canadian province of Manitoba
  Interventions: Diagnostic Test: Babesia NAT

INTERVENTIONS:
Diagnostic Test: Babesia NAT — Blood donors will be tested with Babesia NAT

SUMMARY:
Babesia is a parasite that can be transmitted from the bite of a tick to an individual. While many some people may not have any symptoms from infection, others may experience anything from flu-like symptoms to joint pain, hemolytic anemia, or jaundice. Should an infected individual donate blood, they could pass the infection to a recipient through their blood donation. In 2018, Canadian Blood Services (CBS) screened blood donations between June and October, and Babesia was found in 0.002% - 0.0007% of donors. This prevalence is slightly less than other areas where Babesia testing is not mandated for blood donors (such as Arizona and Oklahoma), and several logs less than areas where Babesia testing is mandated for blood donations. Based on these data, a later Canadian Babesia case, and risk modelling by CBS, a risk-based decision-making (RBDM) process was initiated. The RBDM strongly emphasizes consistent monitoring and frequent testing for Babesia among Canadian blood donors. This proactive strategy is aimed at minimizing the risk of Babesia transmission through donated blood. This study will span five years and examine the prevalence of Babesia, other tick-borne diseases (such as Anaplasma and Powassan virus), and other emerging pathogens which may impact the blood supply.

DETAILED DESCRIPTION:
Overview: This multi-year study will span five years and will examine the prevalence of tick-borne and emerging pathogens that may impact the safety of the blood supply. An overview of the timeline of the study is attached as Figure 1. This study will have a direct impact on the screening of blood donations for infectious disease and will be used to implement evidence-based policy decisions for screening recommendations.

Blood donation: Whole blood donors donating blood in the identified geographic regions will arrive at the Donation Center as routine. When they arrive, they will be asked to read: (1) "What happens to your donation" pamphlet , which describes that "parts of your donation may be used… for quality assurance purposes, evaluating the blood supply process and product improvement testing;" (2) "What you must know to donate blood" pamphlet , which indicates that "other tests may be done on some donations as required", and that "you will be informed of unusual results from any of the tests that we perform;" and (3) the "Privacy Notice to Blood Donors, Stem Cell Registry Participants and for Canadian Blood Services' Cord Blood Bank" (routine). Only donors who are donating blood as part of their routine self-driven blood donation will be included in the study, participants will not be contacted to come in for blood donation for the purposes of this study. Samples will be collected as part of a normal blood donation. A diversion pouch is routinely collected during each donation. Retention samples (routine) and lysis tubes (study) will be filled on-site at collections from the diversion pouch. Priority will be given to all routine collections from the diversion pouch prior to lysis tube collection. No additional volume will be collected from donors for this study.

Routine Testing: All pre-release testing will be completed as normal, and products will be released into inventory prior to any study testing. Testing performed as part of this surveillance project (Babesia, Anaplasma, etc.) are not considered release tests, and therefore will not affect the available blood supply, nor delay release of any blood products.

Study Testing: Following collection of retention sample and lysis tube, samples will be sent to Ottawa lab for labelling and storage. Samples will be batch tested either in-house with CBS, or by the American Red Cross (ARC). Confirmatory testing or other specialized testing for positive samples may be performed at the National Microbiology Laboratory. Lysis samples will be stored up to one year from time of collection, and residual samples will be stored up to 5 years from time of collection for all samples collected as part of this study to allow for additional markers to be tested as needed..

Result Reporting: All positive results will be communicated to the donor via the CBS Medical Office (letter) and by the CBS Medical Officer (phone call) to explain risk factor data and notify of indefinite deferral. Provincial MOHs will be notified of positive results in accordance with provincial communicable disease reporting. If a positive is found, transfusable components associated with that donation will be recalled.

Data Access and Data Analysis: Data will be uploaded to CBS Data Storage and linked with the donation number. Donation number is not identifiable outside of access to CBS eProgesa. Epidemiology and Surveillance Team will link data on secure CBS server (data stored only on servers and database systems, not on laptops). All data will be retrieved from CBS records and merged with the surveillance testing data. Aggregate non-identifiable data will be presented and published for knowledge translation. Study data will be shared in the Surveillance Report and ongoing study information will be added to the website. Data will be stored for 10 years and will be used to affect evidence-based policy decisions on emerging pathogens in the Canadian blood supply.

ELIGIBILITY:
Inclusion Criteria:

* all whole blood donors giving blood in Manitoba during the study period

Exclusion Criteria:

* individuals not eligible to donate blood

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Only blood donors will be included in this study. Minimum age for whole blood donation is 17 years and there is no maximum age limit. Eligibility for donation requires donors to be healthy at time of collection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of Babesia in Canadian Blood Donors | Anticipated July 2 2024 to Oct 25 2024
  All whole blood donors in Manitoba will be tested for Babesia

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Charlton, PhD, Study Chair — Canadian Blood Services; Steven Drews, PhD, Study Director — Microbiology, Donation Policy And Studies, Canadian Blood Services; Mindy Goldman, MD, Principal Investigator — Canadian Blood Services

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared, individual data will not be shared with outside researchers